CLINICAL TRIAL: NCT04310670
Title: Role of Integrated Treatment in Patients With Functional Neurological Disorder
Brief Title: Integrated Treatment in FND (Functional Neurological Disorders)
Acronym: FND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, Professor, Neuromed IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FND integrated treatment
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Functional Neurological Disorder
Keywords: FND; physiotherapy; psychotherapy; non-invasive brain stimulation
MeSH Terms: conditions — Conversion Disorder | interventions — Psychotherapy; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with FND (Experimental): Diagnosis of Functional Neurological Disorder of movement clinically established according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria
  Interventions: Other: Psychotherapy; Behavioral: Physiotherapy; Other: Non-Invasive Brain Stimulation (NIBS)

INTERVENTIONS:
Other: Psychotherapy — The patient will be treated according to Lacanian psychoanalytic ethics, which allows to adequately respond to the patient's request for healing but who at the same time does not ignore the progress of scientific research in the neurological field
Behavioral: Physiotherapy — Physiotherapy treatment will be articulated through the use of techniques designed to qualify the functionality of the subject divided by symptom: weakness, dystonic attitudes of the limbs, walking disorders, tremor.
Other: Non-Invasive Brain Stimulation (NIBS) — Diversified transcranial electrical maneuver protocols with an "on-line" or "off-line" approach may be applied for therapeutic purposes. This will include: transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), random noise stimulation (tRNS).

SUMMARY:
The project will investigate the effectiveness of patient-centered integrated treatment.

The correlations between physiotherapy indices, non-invasive brain stimulation, connectivity and psychological support will be analyzed.

DETAILED DESCRIPTION:
At the time of recruitment (T0) a multidimensional evaluation will be performed consisting of clinical, neuropsychological, neurophysiological, MRI, data obtained from peripheral blood sampling (10ml). After completing the program (12 weeks), the effect will be assessed according to objectives (T1). The study will also include a follow-up evaluation after 6 months (T2) and 12 months (T3) from the beginning of the treatment to evaluate the persistence of the beneficial effects after some time.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Diagnosis of Functional Neurological Disorder of movement clinically established according to DSM-5 criteria
* Age between 18 and 65 years (inclusive)
* Ability to participate in the study protocol

Exclusion Criteria:

* Inability to provide written informed consent
* Pregnant women
* In case of use of non-invasive brain stimulation techniques: the subjects must not present any of the contraindications specific to this method (for further specifications see the "Methods" and the "Stimulation Evaluation Questionnaire" attached to this proposal)
* Presence of unstable clinical conditions or infections
* In the case of the use of non-invasive brain stimulation techniques: concomitant use of drugs that can alter the transmission and synaptic plasticity (cannabinoids, L-dopa, antiepileptics, nicotine, baclofen, Selective Serotonin Reuptake Inhibitors (SSRI), botulinum toxin)
* Inability to support physiotherapy or psychotherapy sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes and improvement in clinical condition | 1-12 months
  the Clinical global impression scale will be used. It is a brief 3-item observer-rated scale that assess severity of illness with assignable scores ranging from 0 to 7 (at every time time point), the global improvement with assignable scores ranging from 0 to 7 (from the second time point), and the efficacy index with assignable scores ranging from 1 to 16 (relationship between therapeutic efficacy and undesirable effects). Higher scores on these scales mean a worse outcome.
Changes in quality of life | 1-12 months
  The Short Form Health Survey 36 (SF-36) will be used. It is a generic, multidimensional tool, consisting of 36 questions that can be divided into 8 scales (Physical functioning, limitations due to physical health, limitations due to emotional problems, energy and fatigue, emotional well-being, social activities, pain, general health perception) expressed as percentage values 0-100%. Higher scores on these scales mean a better quality of life.
Changes in executive functions and attention - step 1 | 1-12 months
  Will be used the Symbol Digit Modalities Test, which measures the processing speed, in the oral version of this test (Nocentini et al., 2006). The assignable performance's scores ranging from 0 to 110. The cut-off for normality in italian population for this oral version was 34.2. Higher scores on these scales mean a better processing speed.
Changes in executive functions and attention - step 2 | 1-12 months
  Stroop test
Changes in neuroplasticity | 1-12 months
  Transcranial Magnetic Stimulation (TMS) will be used to evaluate the change of neuronal plasticity in a subgroup of patients who will not present contraindications to the method. The TMS uses short-lived magnetic fields and high intensity applied at the scalp level to activate the neurons of a small region of the cerebral cortex through an electromagnetic induction. When these impulses are applied repeatedly, it is possible to induce plastic modification of cortical excitability. Any increase or decrease in amplitude, which persists after the end of TMS repetitive stimulation, indicates that there have been changes in the cortical, long term potentiation (LTP) or depression (LTD).
Evaluation of genetic polymorphisms | 1-12 months
  A blood sample (10 ml) will be collected to investigate whether genetic polymorphisms related to patients' neuronal plasticity can be related to the response to the protocol.

SECONDARY OUTCOMES:
Changes in behavioral aspects - step 1 | 1-12 months
  State-Trait Anxiety Inventory-Form Y (STAI-Y). The STAI-Y is a self-report questionnaire consisting of two 20-item scales providing separate measures of state and trait anxiety, on a 4-point Likert scale, with scores ranges from 20 to 80, with higher scores indicating more severe outcome.
Changes in behavioral aspects - step 2 | 1-12 months
  Beck Depression Inventory - Second Edition (BDI-II). BDI-II is a self-report questionnaire consisting of 21-item self-report scale designed to measure the severity of depressive symptoms, on a 4-point Likert scale, with scores ranges from 0 to 63, with higher scores indicating more severe outcome.
Changes in behavioral aspects - step 3 | 1-12 months
  Toronto Alexithymia Scale (TAS-20). TAS-20 is a self-report questionnaire scale designed to measure alexithymia, on a 5-point Likert scale, with scores ranges from 20 to 100, with higher scores indicating more severe outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, Principal Investigator — IRCCS Neuromed
Locations (1):
- I.R.C.C.S. NEUROMED Istituto Neurologico Mediterraneo, Pozzilli, Isernia, Italy

REFERENCES:
- [Result] Galli S, Bereau M, Magnin E, Moulin T, Aybek S. Functional movement disorders. Rev Neurol (Paris). 2020 May;176(4):244-251. doi: 10.1016/j.neurol.2019.08.007. Epub 2019 Oct 9. PMID 31606137
- [Result] O'Neal MA, Baslet G. Treatment for Patients With a Functional Neurological Disorder (Conversion Disorder): An Integrated Approach. Am J Psychiatry. 2018 Apr 1;175(4):307-314. doi: 10.1176/appi.ajp.2017.17040450. No abstract available. PMID 29606068